CLINICAL TRIAL: NCT03560024
Title: The Effect of PACAP27 on the Extra- and Intracerebral Arteries Assessed by MRA on Healthy Volunteers
Brief Title: The Effect of PACAP27 on the Extra- and Intracerebral Arteries Assessed by Magnetic Resonance Angiography (MRA) on Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, Principal Investigator, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-18016693
Record Dates: First submitted 2018-06-01; First posted 2018-06-18 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Intervention Model Description: 18 healthy volunteers will receive PACAP27 or placebo. All Data will also be analyses blinded.
Who Masked: Participant, Investigator
Masking Description: Randomized, double-blind placebo-controlled design in healthy volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACAP27 (Active Comparator): 12 healthy volunteers will receive PACAP27 (10 picomole/kg/min) over 20 min
  Interventions: Other: PACAP27
- Placebo (Placebo Comparator): 6 healthy volunteers will receive placebo (Saline) over 20 min
  Interventions: Other: Placebo

INTERVENTIONS:
Other: PACAP27 — PACAP27 is vasodilator of cerebral vessels
  Arms: PACAP27
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
Studying Pituitary adenylate cyclase-activating peptide 27 (PACAP27) effects on extra- and intracerebral arteries assessed by MRA on healthy volunteers.

DETAILED DESCRIPTION:
PACAP neuropeptide, which belongs to the vasoactive intestinal polypeptide (VIP)/glucagon/secretin family. PACAP exists in two forms: Studying Pituitary adenylate cyclase-activating peptide 38 (PACAP38), which consists of 38 amino acids and PACAP27 which contains 27 amino acids at its N-terminus. PACAP38 is implicated in migraine pathophysiology however PACAP27 is not studied well. Therefore, the investigators will study PACAP27's effect on extra- and intracerebral arteries assessed by MRA on healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-50
* 50-100 kg

Exclusion Criteria:

* Tension type headache more than 5 dag /month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the half-life for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease
* Primary relatives with current or previous migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Dilation of extra- and intracerebral arteries | 0-290 min
  A single-slab 3D time-of-flight (3D TOF) MRA of extra- and intracranial arteries will be acquired as described in previous studies (Amin et al., 2013, 2014). MRA data will be analyzed by LKEB-MRA vessel wall analysis software program. We will measure the circumference of vessels in millimeter in five predefined time points (0, 20, 110, 200 and 290 min)

SECONDARY OUTCOMES:
Headache | 0 to 24 hours
  Headache intensity (Visual analog scale 0-10), characteristics, location and migraine associated symptoms will be recorded in questionnaire at hospital (6 hours) and post hospital (18 hours). In hospital phase, headache questionnaire will be filled every 30 min and post hospital every hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No